CLINICAL TRIAL: NCT05395455
Title: Effect of Non-surgical Periodontal Treatment on Gingival Crevicular Fluid, Salivary and Serum Interleukin-26 Levels in Stage III Grade B and C Periodontitis
Brief Title: Gingival Crevicular Fluid, Salivary, and Serum Biomarkers Levels in Periodontal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAG-C-DRP-241018-0575
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Periodontal Health; Periodontitis
Keywords: periodontitis; periodontal treatment
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Periodontally Healthy (No Intervention): Systemically and periodontally healthy
- Stage III Grade B Periodontitis (Active Comparator): The patients were subjected to quadrant-wise full-mouth subgingival scaling and root planing under local anesthesia. The entire non-surgical periodontal treatment of periodontitis groups was completed in a total of 4 sessions in two weeks.
  Interventions: Procedure: Non-surgical periodontal treatment
- Stage III Grade C Periodontitis (Active Comparator): The patients were subjected to quadrant-wise full-mouth subgingival scaling and root planing under local anesthesia. The entire non-surgical periodontal treatment of periodontitis groups was completed in a total of 4 sessions in two weeks.
  Interventions: Procedure: Non-surgical periodontal treatment

INTERVENTIONS:
Procedure: Non-surgical periodontal treatment — Treatment of patients with periodontitis was performed scaling and root planing by using manual and ultrasonic instruments.
  Arms: Stage III Grade B Periodontitis; Stage III Grade C Periodontitis

SUMMARY:
The present study aimed to assess the effect of non-surgical periodontal treatment on gingival crevicular fluid (GCF), saliva, and serum IL-26, IL-6, and IL-10 levels in stage III grade B periodontitis (SIII-GB-P) and C periodontitis (SIII-GC-P) patients. 25 periodontally healthy, 25 SIII-GB-P, and 25 SIII-GC-P participants were enrolled. At baseline, GCF, saliva, and serum samples were collected and the whole mouth clinical periodontal parameters were recorded. Periodontitis patients received non-surgical periodontal treatment (NSPT). Clinical parameters and samples were re-collected at 1 and 3 months after NSPT. GCF, saliva, and serum IL-26, IL-6, and IL-10 were analyzed by ELISA. Data were analyzed using appropriate statistical tests.

DETAILED DESCRIPTION:
Periodontitis is an inflammatory process that can result in tooth loss by destroying teeth-supporting tissues. Interleukin (IL) 26, is one of the recent members of the IL-10 cytokine family. The elevated level of IL-26 expression is associated with inflammatory disorders.

IL-6, a pro-inflammatory cytokine and is one of the important molecules in the regulation of inflammatory immune responses in periodontitis. IL-10, an anti-inflammatory cytokine, affects monocytes and macrophages and their immune mediator release.

This study is the first controlled clinical study that examines the levels of IL-26 in GCF, saliva, and serum in two different periodontitis, and evaluates the situation before and after the treatment. The first hypothesis of this study GCF, salivary, and serum IL-26 and IL-6 levels will be high and GCF, salivary and serum IL-10 will be low in periodontitis groups, in contrast to the periodontal health the second hypothesis of this study is that after periodontal treatment, GCF, saliva, and serum IL-26 and IL-6 will decrease and GCF, saliva, and serum IL-10 will increase.

Based on these hypotheses, the aim of the study is; to compare the levels of IL-26, IL-6, and IL-10 in GCF, saliva, and serum of healthy controls, SIII-GB-P, and SIII-GC-P subjects and to evaluate the effect of periodontal treatment.

A total of 75 systemically healthy patients; 25 periodontally healthy, 25 SIII-GB-P, and 25 SIII-GC-P were included in this study. The clinical periodontal examination, including measurement of probing depth (PD), clinical attachment level (CAL), bleeding on probing (BOP), gingival index (GI), and plaque index (PI) was performed at 6 sites per tooth, except the third molars. The presence of alveolar bone loss was assessed on the digital panoramic radiograph in each participant, which was supplemented with periapical radiographs if necessary.

The periodontal status of each patient was evaluated by a single calibrated periodontist with a manual probe. The diagnosis of periodontitis or periodontally health was determined according to the 2017 World Workshop on Classification of Periodontal and Peri-Implant Diseases and Conditions. Periodontally healthy individuals (n=25) in the control group had no sites with PD >3 mm and CAL >2 mm and also no radiographic evidence of alveolar bone loss. BOP was <10% in the whole mouth and exhibited no history of periodontitis. The periodontitis stage III patients had a minimum of 3 teeth apart from the first molars and incisors showing CAL ≥5 mm and PD ≥6 mm and showed no>4 teeth loss caused by periodontitis. The radiographic bone loss extends from coronal to middle third or beyond. Radiographic bone loss was determined from the tooth showing the most severe bone loss as a percentage of root length. If the values of bone loss %/age were between 0.25 and 1.0, the patients were assigned to grade B (n=25). If higher than 1.0, the patients were assigned to grade C (n=25).

Treatment The periodontitis patients received conventional scaling and root planning (SRP) under local anesthesia in a total of 4 sessions in two weeks. SRP was performed by the same periodontist using ultrasonic inserts and manual periodontal curettes. Re-evaluations were performed at 1 and 3 months following the completion of the treatment.

GCF, Saliva and Serum Sampling Filter paper strips were used to collect GCF samples. In the healthy control group, GCF was collected from the interproximal sites of single-rooted and multiple rooted teeth from each quadrant. GCF was collected from the sites with PD ≥ 6 mm and radiographic bone loss in periodontitis groups. Selected sites were isolated with cotton rolls. The paper strip was removed after 30 sec after inserting the periodontal pocket. A total of 5 mL of unstimulated whole saliva was collected by the passive drool method in the morning. The saliva was collected over a period of 5 minutes with instructions to pool saliva on the floor of the mouth and passively drool it into a sterile glass beaker and samples are immediately transferred to a 2 mL polypropylene tube. A total of 5 mL of blood was collected from the antecubital fossa by venepuncture method. Serum was isolated from the blood by centrifuging at 5000 rpm for 10 minutes followed by its rapid transfer to a sterile polypropylene tube. All the samples were stored at -80°C.

Biomarker Immunoassays GCF, saliva, and serum samples were thawed on ice. The saliva samples were centrifuged at 5.000 rpm for 15 minutes at room temperature, and supernatants were immediately used for assays. GCF, serum, and salivary samples of IL-26, IL-10, and IL-6 were measured by ELISA using commercial kits.

Statistical Analysis All statistical analyses were carried out with the standard statistical software package. For the intra-group comparisons, if the data were not normally disturbed, the Friedman test and the Dunn test with the Bonferroni correction were used to analyze the change between baseline and 1 month and 3 months after treatment. For inter-group comparisons, the Mann-Whitney U test was performed. The Spearman's rank correlation test was used to detect the correlations of biochemical parameters with clinical parameters and each other in periodontitis group before and after treatment. All tests were performed at a significance level of p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy and non-smoker individuals
* having ≥20 teeth present (except third molars)
* individuals with periodontally healthy, stage III grade B and C periodontitis diagnoses

Exclusion Criteria:

* having any diagnosed medical disorders
* usage of antibiotics, non-steroidal anti-inflammatory drugs, and immunosuppressive agents within the past 6 months
* having any non-inflammatory destructive periodontal disease
* non-surgical/surgical periodontal therapy received in the past year
* pregnant/ lactating/ postmenopausal females

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
GCF IL-26 level (ng/ml) | Baseline to 1 month and 3 months after treatment
  Change in GCF IL-26 levels from baseline to 1 month and 3 months after treatment
GCF IL-6 level (ng/ml) | Baseline to 1 month and 3 months after treatment
  Change in GCF IL-6 levels from baseline to 1 month and 3 months after treatment
GCF IL-10 level (ng/ml) | Baseline to 1 month and 3 months after treatment
  Change in GCF IL-10 levels from baseline to 1 month and 3 months after treatment

SECONDARY OUTCOMES:
Saliva IL-26 level (ng/ml) | Baseline to 1 month and 3 months after treatment
  Change in saliva IL-26 levels from baseline to 1 month and 3 months after treatment
Saliva IL-6 level (ng/ml) | Baseline to 1 month and 3 months after treatment
  Change in saliva IL-6 levels from baseline to 1 month and 3 months after treatment
Saliva IL-10 level (ng/ml) | Baseline to 1 month and 3 months after treatment
  Change in saliva IL-6 levels from baseline to 1 month and 3 months after treatment
Serum IL-26 level (ng/ml) | Baseline to 1 month and 3 months after treatment
  Change in serum IL-26 levels from baseline to 1 month and 3 months after treatment
Serum IL-6 level (ng/ml) | Baseline to 1 month and 3 months after treatment
  Change in serum IL-6 levels from baseline to 1 month and 3 months after treatment
Serum IL-10 level (ng/ml) | Baseline to 1 month and 3 months after treatment
  Change in serum IL-10 levels from baseline to 1 month and 3 months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Hatice Selin Yıldırım, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided